CLINICAL TRIAL: NCT04435314
Title: Prospective, Randomized, Double-blind, Parallel, Placebo Controlled Study to Evaluate the Safety and Efficacy of Nitazoxanide 600 mg Three Times a Day for Post Exposure Prophylaxis of COVID-19 in Subjects From Vulnerable Communities
Brief Title: Efficacy and Safety of Nitazoxanide for Post Exposure Prophylaxis of COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's strategic decision
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NITFQM0620OR
Record Dates: First submitted 2020-06-08; First posted 2020-06-17 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: covid19
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either nitazoxanide (n=100) or placebo (n=100)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitazoxanide (Experimental): Subjects will receive nitazonanide 600 mg TID.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Subjects will receive placebo TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Subjects will receive nitazonanide 600 mg TID for 7 days
  Other Names: Viranitta
  Arms: nitazoxanide
Drug: Placebo — Subjects will receive placebo TID for 7 days.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the drug nitazoxanide 600 mg, administered three times a day, in relation to placebo in preventing the development of COVID-19 in subjects from vulnerable communities that had direct contact with patients diagnosed with the disease.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of the drug nitazoxanide 600 mg, administered three times a day, in relation to placebo in preventing the development of COVID-19 in subjects from vulnerable communities that had direct contact with patients diagnosed with the disease.

Subjects that PCR is negative after having direct contact with symptomatic subjects and diagnosed with COVID-19 (PCR positive) will be randomized to receive Nitazoxanide TID or placebo TID for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from patient or legal representative.
* Subject of both genders (male and female not pregnant and not breastfeeding) aged 18 years or over;
* Subject that lives in a vulnerable community;
* Subject that were in direct contact with confirmed cases of SARS-CoV-2 infection, as they live or work directly with index patients;
* Not showing symptoms compatible with COVID-19 and and that do not have a positive RT-PCR test in a nasopharyngeal swab sample before randomization;
* Participant capable of understanding and fulfilling all activities planned for the study;
* In use of an acceptable method of contraception throughout the study.

Exclusion Criteria:

* Participating in another RCT in the past 12 months;
* Positive PCR result for COVID-19 during screening;
* History of infection confirmed by SARS-CoV-2;
* Present symptoms suggestive of SARS-CoV-2 infection;
* Presence of comorbidities, which have a contraindication to the use of the study product, not being restricted to:

  * HIV or HTLV virus infection;
  * Chronic hepatitis C (HCV) treated with direct antiviral drugs;
  * Liver failure;
  * Severe renal failure, including dialysis;
* Present hypersensitivity to the study product (nitazoxanide), as well as to related compounds;
* Concomitant administration of drugs that may interact with the product under study (nitazoxanide);
* Participants who underwent treatment with antivirals and / or antiparasitic drugs in the last 30 days;
* Subject in antineoplastic treatment with chemotherapy or radiation therapy;
* Subject with severe autoimmune diseases in immunosuppression;
* Transplanted participants;
* Pregnant or lactating women;
* Any other clinical condition that is deemed by the Investigator to be an imminent risk to the health and life of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with laboratory-confirmed COVID-19 identified after start of treatment and before the end of the study | 28 days
  PCR will be done to evaluate infection

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Number of participants with treatment-related adverse events
The proportion of subjects with symptomatic laboratory-confirmed COVID-19 identified after start of treatment and before the end of the study | 28 days
  Symptomatic PCR positive subjects
The proportion of subjects with asymptomatic laboratory-confirmed COVID identified after the start of treatment and before the end of the study | 28 days
  Asymptomatic PCR will be done to evaluate infection
Treatment adherence | 7 days
  Subject adherence to treatment will be assessed through study diary record
Disease complication | 28 days
  Proportion of patients with severe condition
Incidence of subjects that underwent unscheduled visit | 28 days
  Proportion of patient that needed undergo an unscheduled visit

CONTACTS AND LOCATIONS:
Overall Officials: Reginaldo Raimundo Fujita, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.